CLINICAL TRIAL: NCT00547105
Title: A Phase II Trial of Erlotinib (Tarceva®) in Combination With Stereotactic Body Radiation Therapy (SBRT) for Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Erlotinib and SBRT in Treating Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCC-0609131; SCCC-042007-003 (Other: UT Southwestern); CDR0000571634 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2018-04

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; stage IIIA non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Radiosurgery

STUDY DESIGN:
Intervention Model Description: This study is a single arm phase II pilot trial. Patients enrolled on the trial will have been receiving or will begin to receive erlotinib at standard doses (150 mg po per day). SBRT will commence within 4 weeks of the initiation of erlotinib. Maintenance erlotinib will continue until disease progression uncontrollable by SBRT, intolerable toxicity, or death.

ARMS (1):
- erlotinib in combination with SBRT (Experimental): Patients enrolled on the trial will have been receiving or will begin to receive erlotinib at standard doses (150 mg po per day). SBRT will commence within 4 weeks of the initiation of erlotinib
  Interventions: Drug: Erlotinib; Radiation: SBRT

INTERVENTIONS:
Drug: Erlotinib — Erlotinib is indicated for the treatment of patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) after failure of at least one prior chemotherapy regimen.
  Other Names: Tarceva
Radiation: SBRT — SBRT is a treatment method to deliver a high dose of radiation to the target, utilizing either a single dose or a small number of fractions with a high degree of precision within the body
  Other Names: stereotactic body radiation therapy

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Giving erlotinib together with stereotactic body radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving erlotinib together with stereotactic body radiation therapy works in treating patients with locally advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the effect of erlotinib and stereotactic body radiotherapy on 6-month progression-free survival of patients with locally advanced or metastatic non-small cell lung cancer.

Secondary

* To describe the actuarial rate of in-field local control and out-of-field disease progression in patients treated with this regimen.
* To evaluate the safety of this regimen in these patients.
* To evaluate overall survival of patients treated with this regimen.
* To evaluate the duration of erlotinib usage and time to initiation of third-line systemic therapy (chemotherapy or biologic agent) in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral erlotinib hydrochloride once daily in the absence of disease progression or unacceptable toxicity. Beginning 1-4 weeks after the initiation of erlotinib hydrochloride, patients undergo stereotactic body radiotherapy.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

1. Patients must have biopsy proven NSCLC that is locally advanced or metastatic.
2. Patients must have had failure of at least one prior chemotherapy regimen.
3. Patients must not have started erlotinib therapy more than 4 weeks prior to the initiation of SBRT.
4. Age ≥ 18 years
5. Patients must have measurable disease at baseline.
6. Patients can have up to only 6 discrete active extracranial lesions (≤3 in the liver and ≤3 in the lung) identified by PET scan and also seen on correlative plain film, CT scan, or MRI within 8 weeks prior to the initiation of SBRT.

   1. For patients who have received prior radiotherapy to the primary site in the lung, residual PET activity is difficult to interpret and will not be considered a site of active disease if the CT appearance is stable or improved over an interval of at least three months
   2. Patients who previously received radiotherapy to the primary site will be ineligible if there is CT evidence of disease progression within the past 3 months.
   3. Patients with previously un-irradiated primary sites will be potentially eligible, but special considerations apply (section 4.3.2).
   4. Up to 2 contiguous vertebral metastases will be considered a single site of disease.
7. Patients must have a KPS >60
8. AST, ALT & Alkaline phosphates must be ≤ 2.5X the upper limit of normal. Total bilirubin must be within the limit of normal.
9. Patients should have adequate bone marrow function as defined by peripheral granulocyte count of ≥1500/mm³.
10. Patients should have adequate renal function (serum creatinine ≤1.5 times the ULN).
11. Females of childbearing potential should have a negative pregnancy test.
12. Patients who would be receiving SBRT for lung tumors who are known or suspected by the treating radiation oncologist to have compromised lung function must have a documented forced expiratory volume in 1 second (FEV1) ≥ 1L.
13. Patients must provide verbal and written informed consent to participate in the study.
14. Total bilirubin: within normal institutional limits

Exclusion Criteria Patients who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Patients who previously received radiotherapy to the primary site with CT evidence of disease progression at the primary site within 3 months following the initial radiotherapy.
2. Patients with either untreated brain metastases or brain metastases treated within the past three months are ineligible
3. Patients with serious, uncontrolled, concurrent infection(s).
4. Significant weight loss (>10%) in the prior 3 months.
5. Because the tolerance dose of SBRT to the gastrointestinal tract is not established, patients with metastatic disease invading the esophagus, stomach, intestines, or mesenteric lymph nodes will not be eligible.
6. Patients with cutaneous metastasis of NSCLC.
7. Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cancers.
8. Patients with more than 6 discrete extra-cranial lesions.
9. Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
10. Unwillingness to participate or inability to comply with the protocol for the duration of the study.
11. Patients who are pregnant. Patients with reproductive capability will need to use adequate contraception during the time of participation in the study.
12. Patients who have had prior EGFR inhibitors.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06-25 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2017-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Timmerman, MD, Study Chair — Simmons Cancer Center
Locations (2):
- United States (2):
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Body Radiation Therapy Combined With Erlotinib: Patients enrolled on the trial will have been receiving or will begin to receive erlotinib at standard doses (150 mg po per day). Stereotactic Body Radiation Therapy (SBRT) will commence within 4 weeks of the initiation of erlotinib
  Erlotinib: Erlotinib is indicated for the treatment of patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) after failure of at least one prior chemotherapy regimen.
  SBRT: SBRT is a treatment method to deliver a high dose of radiation to the target, utilizing either a single dose or a small number of fractions with a high degree of precision within the body
Period: Overall Study
Arm/Group | Stereotactic Body Radiation Therapy Combined With Erlotinib
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- SBRT in Combination With Erlotinib: Patients enrolled on the trial will have been receiving or will begin to receive erlotinib at standard doses (150 mg po per day). SBRT will commence within 4 weeks of the initiation of erlotinib
  Erlotinib: Erlotinib is indicated for the treatment of patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) after failure of at least one prior chemotherapy regimen.
  SBRT: SBRT is a treatment method to deliver a high dose of radiation to the target, utilizing either a single dose or a small number of fractions with a high degree of precision within the body
Arm/Group | SBRT in Combination With Erlotinib
Number analyzed (Participants) | 24
Age, Continuous [Median (Full Range); unit: years] | 67 [56 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression-Free Survival
Description: For liver lesions treated with SBRT, RECIST (Response Evaluation Criteria in Solid Tumors) criteria will be used for evaluation of progression. Progression (PD) is at least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Evaluation of lung lesions at any time after SBRT is difficult in view of the expected fibrotic reaction. Bone lesions seen only on PET are also not well scored by RECIST criteria and will not be evaluated in that manner. In this study progressive disease (PD) will be defined as residual increased metabolic PET scan in combination with expanded parenchymal opacity that retains mass-like discrete borders and extends outside the volume of lung that received at least 18 Gy.
Time Frame: 6 months
Population: Twenty-four patients with stage IV Non-small-Cell Lung Caner with six or fewer sites of disease after progressing through first-line or subsequent systemic therapy were enrolled on the study.
Measure: Number; unit: percentage of participants
Groups:
- SBRT Combined With Erlotinib: Patients enrolled on the trial will have been receiving or will begin to receive erlotinib at standard doses (150 mg po per day). SBRT will commence within 4 weeks of the initiation of erlotinib
  Erlotinib: Erlotinib is indicated for the treatment of patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) after failure of at least one prior chemotherapy regimen.
  SBRT: SBRT is a treatment method to deliver a high dose of radiation to the target, utilizing either a single dose or a small number of fractions with a high degree of precision within the body
Arm/Group | SBRT Combined With Erlotinib
Number analyzed (Participants) | 24
percentage of participants | 69

2. Secondary Outcome: In-field Local Control
Description: In-field local control is defined as number of treated lesions that did not grow in size or increase in metabolic activity.
Time Frame: 9 months
Population: 21 out of 24 patients were evaluable with baseline and minimum 3-month follow-up CT based imaging. The other three patients died or had not otherwise reached this window for evaluation.
Measure: Count of Units; unit: lesions treated with SBRT
Units Other Than Participants: lesions treated with SBRT
Arm/Group | SBRT Combined With Erlotinib
Number analyzed (Participants) | 21
Number analyzed (lesions treated with SBRT) | 47
lesions treated with SBRT | 44

3. Secondary Outcome: Number of Participants Without Serious Adverse Events Related to Radiation
Description: Common Terminology Criteria for Adverse Events v4.03 (CTCAE) is used as the standard classification and severity grading scale for adverse events
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT Combined With Erlotinib
Number analyzed (Participants) | 24
Participants | 22

4. Secondary Outcome: Overall Survival
Description: evaluate overall survival after SBRT in combination with erlotinib
Time Frame: up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | SBRT Combined With Erlotinib
Number analyzed (Participants) | 24
months | 20.4 [3 to 60]

5. Secondary Outcome: Duration of Erlotinib Use and Time to Initiation of Third-line Systemic Therapy
Description: To evaluate the duration of erlotinib usage and time to initiation of third line systemic agent (chemotherapy or biologic agent)
Time Frame: 3 years
Measure: Median (Full Range); unit: days
Arm/Group | SBRT Combined With Erlotinib
Number analyzed (Participants) | 24
days | 183 [24 to 847]

6. Secondary Outcome: Out-of-field Disease Progression
Description: Number of Participants with Disease Progression Outside the Radiation treated field at 9 Months
Time Frame: 9 months
Population: The other three patients died or had not otherwise reached this window for evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT Combined With Erlotinib
Number analyzed (Participants) | 21
Participants | 10

7. Secondary Outcome: Progression-free Survival
Description: as for outcome 1
Time Frame: up to 5 years
Measure: Median (Full Range); unit: months
Arm/Group | SBRT Combined With Erlotinib
Number analyzed (Participants) | 24
months | 14.7 [2 to 60]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | SBRT Combined With Erlotinib
All-Cause Mortality (participants affected / at risk) | 13/24
Serious Adverse Events (participants affected / at risk) | 5/24
Other Adverse Events (participants affected / at risk) | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT Combined With Erlotinib (N=24)
Pneumonitis grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) — definitely related to radiation
diarrhea grade 4 (Gastrointestinal disorders) | 3 (3) — definitely related to erlotinib
spinal fraction grade 3 (Injury, poisoning and procedural complications) | 1 (1) — back pain definitely related to radiation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes